CLINICAL TRIAL: NCT02577172
Title: Testicular Cancer and Aerobic and Strength Training - a Randomized Controlled National Phase II Study
Brief Title: Testicular Cancer and Aerobic and Strength Training
Acronym: TAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected events
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Lene Thorsen, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REK - 2014/1169
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Testicular Neoplasms
Keywords: Testicular cancer; Physical Exercise; Chemotherapy
MeSH Terms: conditions — Testicular Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Aerobic- and Strength Training program
  Interventions: Behavioral: Exercise group
- Control group (Active Comparator): One lifestyle counseling session
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Exercise group — The intervention will be conducted during chemotherapy and tailored for each patient. The program will include 1) weight bearing aerobic exercises to maintain the oxygen transport and thereby reduce the decline in VO2max during chemotherapy and 2) strength training exercises to maintain muscle mass and muscle strength. The intervention will last for 9 or 12 weeks, depending on the number of BEP/EP cycles received. The program will consist of two-three one-hour exercise sessions per week, of which most supervised by a personal trainer. The intensity of each exercise sessions will varies from easy (warm-up: 60-70 % of peak heart rate) to moderate/high (between aerobic intervals 60-70% of peak heart rate and during aerobic intervals 85-95 %).
  Arms: Exercise group
Behavioral: Control group — The control group will receive one individual lifestyle counseling session during the first chemotherapy cycle and can perform all activities that they have planned to do during chemotherapy.
  Arms: Control group

SUMMARY:
The present study examine the effects of an aerobic and strength training program on cardiorespiratory fitness in testicular cancer (TC) patients during chemotherapy. Half of the participants will receive the exercise program and the other half will receive one individual lifestyle counseling session. The investigators hypothesize that TC patients in the exercise group will have less reduction in cardiorespiratory fitness during chemotherapy treatment compared to patients in the control group.

DETAILED DESCRIPTION:
Testicular cancer (TC) patients receiving chemotherapy often experience troublesome side-effects during and after treatment. Both aerobic and strength exercise have showed beneficial effects on side-effects during and after treatment in other cancer diagnosis. Knowledge of the effects of physical exercise during and after chemotherapy in TC patients is insufficient and studies are needed. The primary aim is to examine the effects of physical exercise on cardiorespiratory fitness in TC patients during chemotherapy. Secondary aims are to examine the effects of physical exercise on other secondary health outcomes during and three and twelve months after chemotherapy.

The present study is a randomized controlled trial comparing a tailored exercise program consisting of aerobic and strength training during chemotherapy to a control group receiving one individual lifestyle counseling session during the first chemotherapy cycle. The TC patients will be included and assessed before the first cycle of chemotherapy and further assigned to either a exercise group or a control group. The intervention will last for 9 or 12 weeks (depending on the number of bleomycin, etoposide, cisplatin (BEP)/etoposide, cisplatin (EP) cycles received) and it will consists of two-three one-hour sessions per week mostly supervised by a personal trainer. All variables will be assessed pre- and post-intervention, and at three and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* testicular cancer with seminoma or non-seminoma
* stage II-IV
* referred to chemotherapy (3-4 BEP (bleomycin, etoposide and cisplatin)-cycles or 4 EP (etoposide and cisplatin) -cycles) with/without retroperitoneal lymph node dissection (RPLND)
* satisfactory Norwegian Language skills
* signed informed consent

Exclusion Criteria:

* severe brain and lung metastasis (reduced lung function)
* heart and lung diseases that contraindicate exercise testing and the supervised exercise program without adjusted actions according to American College of Sports Medicine (ACSM)'s guidelines)
* physical and mental conditions of a severity that complicates the ability for exercise testing and the supervised exercise program

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
VO2peak (directly by modified Balke protocol on a treadmill) | Pre-intervention (week 0) to post-intervention (week 10/13)
  Differences in change in VO2peak from pre- to post-intervention between the exercise group and the control group.

SECONDARY OUTCOMES:
VO2peak (directly by modified Balke protocol on a treadmill) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in VO2peak from pre-post-intervention to three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of reduced VO2peak at 12 months follow-up in all participants.
Spirometry | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in pulmonary function (lung capacity, lung volume, diffusion capacity) from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group.
One-repetition maximum muscle strength test (1RM) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in muscle strength from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group.
Dual-energy X-ray absorptiometry (DXA) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in lean body mass and fat mass from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of unhealthy body composition at 12 months follow-up in all participants.
Body mass index (BMI) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in BMI from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of unhealthy BMI at 12 months follow-up in all participants.
Hip- and Waist circumferences | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in hip- and waist circumferences from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group.
Godin Leisure Time Exercise Questionnaire (GLTEQ) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in physical exercise from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of being inactive at 12 months follow-up in all participants.
Sick leave and Work Ability Index (WAI) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in work ability and sick leave from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of reduced work ability at 12 months follow-up in all participants.
The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C-30 | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in health related quality of life (HRQOL) from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of having reduced HRQOL at 12 months follow-up in all participants.
Fatigue questionnaire | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in fatigue from pre- to post-intervention and at three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of having fatigue at 12 months follow-up in all participants.
Hospital and Anxiety and Depression Scale (HADS) | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in anxiety and depression from pre- to post-intervention and to three and 12 months follow-ups between the exercise group and the control group. Examine potential prognostic factors of having anxiety and depression at 12 months follow-up in all participants.
Markers for inflammation, endothelia dysfunction, thrombosis and cardiovascular diseases and cisplatin | Pre-intervention (week 0) to post-intervention (week 10/13) and at three and 12 months follow-ups
  Differences in change in blood tests from pre- to post intervention and at three and 12 months follow-up in the exercise group and the control group. Examine potential risk factors for endothelia dysfunction, activated coagulation and thrombosis and cardiovascular diseases (metabolic syndrome) at 12 months follow-up in all participants.
Safety and tolerability | Pre-intervention (week 0) to post-intervention (week 10/13)
  Number of participants with adverse events during the exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thorsen, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Thorsen L, Haugnes HS, Fossa SD, Brydoy M, Tandstad T, Wisloff T, Gjerset GM, Edvardsen E, Larsen KO, Sandset PM, Henriksson CE, Raastad T, Negaard HFS. Thromboembolic events after high-intensity training during cisplatin-based chemotherapy for testicular cancer: Case reports and review of the literature. Int J Cancer. 2020 Dec 1;147(11):3189-3198. doi: 10.1002/ijc.33151. Epub 2020 Jul 1. PMID 32525564